CLINICAL TRIAL: NCT07189013
Title: Assessing Patient Preference for Infusion Systems (Electronic vs. Mechanical)
Brief Title: Assessing Patient Preference for Infusion Systems
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KORU Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KORU0001
Record Dates: First submitted 2025-08-28; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Primary Immunodeficiencies (PID); Secondary Immunodeficiencies (SID)
Keywords: electronic infusion system; mechanical infusion system; immunodeficiency; subcutaneous immunoglobulin administration
MeSH Terms: conditions — Immunologic Deficiency Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Experienced electronic pump users (Experimental): Patients with earlier experience on electronic infusion pumps. They will use the mechanical infusion pump for three months' period.
  Interventions: Device: Mechanical infusion pump

INTERVENTIONS:
Device: Mechanical infusion pump — Patients with earlier experience on electronic infusion pumps will crossover to the mechanical infusion pump for three month's period
  Other Names: Freedom60 Infusion Pump

SUMMARY:
This crossover study evaluates patient experiences and preferences between mechanical and electrical infusion pumps for subcutaneous immunoglobulin (SCIg) therapy. The Freedom Integrated Infusion System (FREEDOM60 and FreedomEdge) are mechanical, portable pumps that require no batteries or electricity and use Precision Flow Rate Tubing™ to control infusion speed. These devices are approved for use in the EU (CE650520).

Approximately 78 adult patients with primary or secondary immunodeficiency will participate. Participants will complete questionnaires assessing ease of training, ease of use, infusion comfort, and overall satisfaction. Patients experienced with electronic pumps will complete two questionnaires: one reflecting their current pump experience and one after trying the mechanical pump.

The primary goal is to determine whether mechanical pumps provide greater patient satisfaction than electrical pumps. Results will inform patient and healthcare professional decision-making regarding pump selection.

DETAILED DESCRIPTION:
Study Objective:

To assess patient preference, ease of training, ease of use, and satisfaction with mechanical versus electrical infusion pump systems.

Subject Population:

Adults with primary or secondary immunodeficiency receiving subcutaneous immunoglobulin therapy, including patients experienced with electronic infusion pumps.

Hypothesis:

Mechanical infusion pumps will provide greater patient satisfaction compared with electrical infusion pumps during SCIg treatment.

Study Assessments / Evaluations:

Experienced electronic pump users will complete two questionnaires: one reflecting their current pump experience and one after trying a mechanical pump. Comparisons will evaluate preference, satisfaction, ease of use, training, infusion comfort, handling, instructions, troubleshooting, and safety.

Number of Subjects:

Approximately 78 patients, completing 130 questionnaires in total.

ELIGIBILITY:
Inclusion Criteria:

* The subject has primary or secondary immunodeficiency or chronic inflammatory demyelinating polyneuropathy and is undergoing IgRT.
* The subject or caregiver is willing and able to provide informed consent.
* The subject has experience using electronic SCIG infusion system (3 months and above).

Exclusion Criteria:

* The subject is participating in another clinical study prior to this study completion.
* The subject has been on IgRT for less than 3 months.
* The subject is less than 18 years old and/or has a legal representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Satisfaction Scores Between Electronic and Mechanical Infusion Pumps Measured on a 5-Point Likert Scale Over 3 Months | Three months
  Participants will first provide a retrospective evaluation of their prior experience with an electronic infusion pump using a 5-point Likert scale (where 1 = worst outcome and 5 = best outcome). They will then crossover to a mechanical infusion pump for 3 months, after which satisfaction will again be assessed on the same scale. The primary outcome is the difference in satisfaction scores between electronic and mechanical pump use.

SECONDARY OUTCOMES:
Change in Ease of Use Scores Between Electronic and Mechanical Infusion Pumps Measured on a 5-Point Likert Scale Over 3 Months | Three months
  Participants will first provide a retrospective evaluation of the ease of use of an electronic infusion pump using a 5-point Likert scale (1 = very difficult to use; 5 = very easy to use). They will then crossover to a mechanical infusion pump for 3 months, after which ease of use will again be assessed on the same scale. The secondary outcome is the difference in ease-of-use scores between electronic and mechanical pump use.
Change in Handling Scores Between Electronic and Mechanical Infusion Pumps Measured on a 5-Point Likert Scale Over 3 Months | Three months
  Participants will first provide a retrospective evaluation of the handling of an electronic infusion pump using a 5-point Likert scale (1 = very difficult to handle; 5 = very easy to handle). They will then crossover to a mechanical infusion pump for 3 months, after which handling will again be assessed on the same scale. The secondary outcome is the difference in handling scores between electronic and mechanical pump use.
Change in Scores for Clarity of Instructions of Use Between Electronic and Mechanical Infusion Pumps Measured on a 5-Point Likert Scale Over 3 Months | Three months
  Participants will first provide a retrospective evaluation of the clarity of instructions of use for an electronic infusion pump using a 5-point Likert scale (1 = very unclear instructions; 5 = very clear instructions). They will then crossover to a mechanical infusion pump for 3 months, after which clarity of instructions of use will again be assessed on the same scale. The secondary outcome is the difference in clarity-of-instructions scores between electronic and mechanical pump use.
Change in Scores for Ability for Troubleshooting Between Electronic and Mechanical Infusion Pumps Measured on a 5-Point Likert Scale Over 3 Months | Three months
  Participants will first provide a retrospective evaluation of the ability for troubleshooting any issues that may arise during the infusion for an electronic infusion pump using a 5-point Likert scale (1 = not at all confident; 5 = very confident). They will then crossover to a mechanical infusion pump for 3 months, after which clarity of instructions of use will again be assessed on the same scale. The secondary outcome is the difference in ability for troubleshooting scores between electronic and mechanical pump use.
Change in Scores for Pain and Discomfort Between Electronic and Mechanical Infusion Pumps Measured on a 5-Point Likert Scale Over 3 Months | Three months
  Participants will first provide a retrospective evaluation of the clarity of instructions of use for an electronic infusion pump using a 5-point Likert scale (1 = extreme pain and discomfort; 5 = no pain and discomfort). They will then crossover to a mechanical infusion pump for 3 months, after which clarity of instructions of use will again be assessed on the same scale. The secondary outcome is the difference in clarity-of-instructions scores between electronic and mechanical pump use.

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No